CLINICAL TRIAL: NCT04688372
Title: Association Between Hospital Case Burden and Mortality Risk Among Patients Hospitalized With COVID-19: A Retrospective Cohort Study of U.S. Hospitals
Brief Title: Hospital COVID-19 Surge and Associated Mortality Risk
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Emory University (Other); Harvard Medical School (HMS and HSDM) (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BD022386
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2020-12

CONDITIONS: Volume Outcome Relationship Among COVID-19 Inpatients in US Hospitals
Keywords: surge; volume; mortality; COVID-19; coronavirus; hospital
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatient encounters with COVID-19 present-on-admission: See Study description above
  Interventions: Other: Surge Index

INTERVENTIONS:
Other: Surge Index — See study description above

SUMMARY:
A retrospective cohort study will be conducted using a large administrative database of U.S. hospitals to understand the volume-outcome relationship among patients hospitalized with COVID-19.

DETAILED DESCRIPTION:
Patients with critical illness and/or respiratory failure tend to display better outcomes at hospitals that manage higher volumes of these patients. However, during a COVID-19 pandemic, this relationship may have been altered by the strain of higher patient volume on resources and personnel. A retrospective cohort study will be conducted using a large administrative database to understand the volume-outcome relationship among patients hospitalized with COVID-19. Understanding the COVID-19 volume-outcome relationship in U.S. hospitals may help identify the optimal care setting and transfer thresholds, and inform triage policies and risk-adjustment.

The Premier Healthcare Database (PHD), an all-payer administrative data repository covering approximately 20% of U.S. hospitalizations from 48 states will be queried for adult (18+ years) in-patient encounters that recorded diagnosis coding for COVID-19 March 1st through August 31st, 2020 at continuously-reporting hospitals. Hospitals with <15 COVID-19 encounters over the study period will be excluded from the primary cohort to preserve statistical reliability.

A surge index will be calculated for each hospital month that incorporates care-complexity-weighted COVID-19 case burden and will be normalized for nominal (2019) bed capacity and non-COVID-19 case burden and will represent the primary covariate. Hospital months will be stratified by the percentile of the surge index (e.g. <50th, 50-75th, 75-90th, 90-95th and ≥95th percentile).

The impact of COVID-19-case burden (surge index) on the risk-adjusted odds ratio (aOR) of mortality (or discharge to hospice) among overall COVID-19 cohorts will be determined using a hierarchical generalized linear mixed model controlling for case-mix, treatment-related, time-varying and other hospital-level factors. Variables will be selected based on their representing "baseline" status upon presentation to the hospital to minimize effect of mediators.

Variables for case mix adjustment: age, gender, race/ethnicity, comorbidity burden, insurance status, admission source and acuity, acute organ failure score and code status present-on-admission, use of pharmacologic agents (remdesivir, corticosteroids, hydroxychloroquine and azithromycin), severity of hypoxia (acute respiratory failure codes, need for non invasive positive pressure ventilation, need for invasive mechanical ventilation), vasopressor use within two days of admission respectively.

Variables for temporal and hospital-level adjustment: hospital teaching status, urbanity, geographic region, bed capacity, hospital proportion of Medicaid/uninsured admissions, proportion of COVID-19 patients intubated within 2 days of admission, hospital's technologic index (stratified by availability of extracorporeal membrane oxygenation, more than one ICU and continuous renal replacement therapy), hospital availability of remdesivir, attending physician to patient ratio, pre-COVID-19 mechanical ventilation volume, proportion of overall admits tested for COVID-19 and admission month (1st vs 2nd wave).

Effect modification by (1st vs. 2nd ) pandemic wave, the previous month's surge index and rate of acute hospital transfers and/or tracheotomies will assessed using interaction terms. Sensitivity analyses will be performed using alternative iterations/strata of the surge index, excluding fewer patients for statistical reliability, models with and without treatment-related variables and using Elixhauser comorbidity index instead of US Centers for Disease Control and Prevention-defined poor prognostic underlying conditions in COVID-19 to test robustness of results. Analyses will be repeated using in-hospital mortality (without reported discharges to hospice). The magnitude of an unmeasured confounder that would be necessary to alter the direction of statistically significant findings will be assessed. More selective subgroups of patients in ICU and mechanical ventilation will not be used as a primary study population given the potentially dynamic nature of admission and intubation criteria over the course of the pandemic and its relationship to volume.

Depending on availability at the time of analysis, an de-identified curated electronic health record-based dataset will be used for clinical validation of select variables in administrative data (e.g. reliability of respiratory failure codes in representing patients requiring high-flow oxygen alone i.e. not non-invasive or invasive mechanical ventilation.)

ELIGIBILITY:
Inclusion Criteria:

* See study description

Exclusion Criteria:

* See study description

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See study description
Sampling Method: Non-Probability Sample
Enrollment: 144116 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality or discharge to hospice | From time of admission to death during the hospitalization or discharge to hospice

SECONDARY OUTCOMES:
In-hospital mortality | From time of admission to death during the hospitalization
  (without reported discharges to hospice)

CONTACTS AND LOCATIONS:
Overall Officials: Sameer S Kadri, MD, MS, Principal Investigator — National Institutes of Health, Clinical
Locations (1):
- National Institutes of Health Clinical Center (primary center conducting large database study), Bethesda, Maryland, United States

REFERENCES:
- [Derived] Kadri SS, Sun J, Lawandi A, Strich JR, Busch LM, Keller M, Babiker A, Yek C, Malik S, Krack J, Dekker JP, Spaulding AB, Ricotta E, Powers JH 3rd, Rhee C, Klompas M, Athale J, Boehmer TK, Gundlapalli AV, Bentley W, Datta SD, Danner RL, Demirkale CY, Warner S. Association Between Caseload Surge and COVID-19 Survival in 558 U.S. Hospitals, March to August 2020. Ann Intern Med. 2021 Sep;174(9):1240-1251. doi: 10.7326/M21-1213. Epub 2021 Jul 6. PMID 34224257